CLINICAL TRIAL: NCT00271206
Title: Progesterone and the Effects of Nicotine
Brief Title: Effect of Progesterone on Smoking Behavior in Male and Female Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0407026935; R01DA014537 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2005-12-28; First posted 2005-12-30 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Tobacco Use Disorder
Keywords: Nicotine Dependence; Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Progesterone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progesterone (Active Comparator): 200 mg to 400mg of progesterone
  Interventions: Drug: Progesterone
- Sugar Pill (Placebo Comparator): Will mirror active medication
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: Progesterone — compared to placebo
  Arms: Progesterone
Drug: sugar pill — Compared to progesterone
  Arms: Sugar Pill

SUMMARY:
Past research on nicotine addiction has shown that changes in estradiol and progesterone hormone levels during menstruation may cause women to respond differently than men to nicotine. The purpose of this study is to examine the effects of progesterone on smoking behavior, nicotine withdrawal symptoms, and the reinforcing effects of smoking in men and women addicted to nicotine.

DETAILED DESCRIPTION:
Nicotine addiction is a serious health problem. Almost 35 million people in the United States try to quit smoking each year, but less than 7 percent are successful. Many smokers report a "high" sensation, followed by a feeling of relaxation. Such positive reinforcement factors, combined with nicotine cravings, make it difficult to stop the use of nicotine products. Past research has suggested that women may experience fewer nicotine cravings and may be less affected by smoking's positive reinforcement factors when compared to men. Fluctuations in levels of the female hormones estradiol and progesterone during menstruation may play a role in determining how women are affected by nicotine. The purpose of this study is to examine the effects of a controlled oral dose of progesterone on smoking behavior, nicotine withdrawal symptoms, and nicotine-related positive reinforcement factors in nicotine dependent males and females.

In this 4-day study, participants will be randomly assigned to receive a daily dose of 200 mg of progesterone, 400 mg of progesterone, or placebo. All participants will abstain from smoking for Days 1 through 3. On Day 4, participants will take part in a smoking session, during which their smoking habits, including the number of puffs, duration of puffs, and number of cigarettes smoked, will be measured. Outcome measurements will include self-reports of cravings; carbon monoxide monitoring; and standardized questionnaires to assess nicotine withdrawal symptoms.

This study has been completed with 35 men and 30 women. With the final women completing in March of 2008. This protocol is complete and has been published.

ELIGIBILITY:
Inclusion Criteria:

* History of smoking 10-25 cigarettes daily for the past 12 months
* Score of at least 5 on the Fagerström Nicotine Tolerance Questionnaire
* Carbon monoxide level greater than 10 ppm
* Body mass index between 19 to 36
* Currently in good health, as determined by medical history, screening examination, and laboratory tests
* If female, regular menstrual cycle every 25 to 35 days
* If female, willing to use non-hormonal contraception throughout the study

Exclusion Criteria:

* Seeking treatment for nicotine dependence
* History of major medical illness, including liver disease; abnormal vaginal bleeding; suspected or known tumors; thrombophlebitis; deep vein thrombosis; pulmonary embolus; clotting or bleeding disorders; heart disease; diabetes; stroke; or other medical conditions that are considered unsafe for study participants by the investigator
* Regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics)
* Recent diagnosis and treatment for Axis I disorders, including major depression, bipolar affective disorder, schizophrenia, or panic disorder
* Currently abusing alcohol or other recreational or prescription drugs
* Current use of any tobacco products other than cigarettes, including smokeless tobacco and nicotine products
* Known allergy to progesterone
* Known allergy to peanuts
* If female, amenorrhea
* Pregnant or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2004-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Smoking topography; measured by carbon monoxide levels and self-report at Day 4 | 4 years anticipated
Nicotine withdrawal symptoms; measured by the Minnesota Nicotine Withdrawal Scale at Day 4 | Anticipated 4 year study

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, PhD, Principal Investigator — Yale University, Department of Psychiatry
Locations (1):
- VA Connecticut Health Care System, New Haven, Connecticut, United States